CLINICAL TRIAL: NCT01808547
Title: A Randomized Double-Masked Study to Compare the Ocular Safety,Tolerability,and Efficacy of ISV-303 to Durasite Vehicle in Cataract Surgery Subjects
Brief Title: Comparison Study of ISV-303 to Durasite Vehicle in Cataract Surgery Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-12-303-004
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Results first posted 2016-07-13 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Ocular Inflammation
MeSH Terms: interventions — bromfenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ISV-303 (Experimental)
  Interventions: Drug: ISV-303
- Durasite Vehicle (Placebo Comparator)
  Interventions: Other: DuraSite Vehicle

INTERVENTIONS:
Drug: ISV-303 — 0.075% bromfenac in DuraSite dosed BID
  Arms: ISV-303
Other: DuraSite Vehicle — DuraSite vehicle dosed BID
  Arms: Durasite Vehicle

SUMMARY:
The purpose of this study is to evaluate the ocular safety, tolerability and efficacy of topical administration of ISV-303 compared with Durasite Vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18 or older scheduled for unilateral cataract surgery with posterior chamber intraocular lens implantation
* If a female is of childbearing potential, the subject must agree to and submit a negative pregnancy test before any protocol-specific procedures are conducted. The subject must use effective contraception for the duration of the study. Post menopausal is defined as having no menses for at least 12 consecutive months
* Signature of the subject on the Informed Consent Form
* Willing to avoid disallowed medications for the duration of the study
* Willing and able to follow all instructions and attend all study visits
* Able to self-administer the IMP (or have a caregiver available to instill all doses of study drugs )
* Additional inclusion criteria also apply

Exclusion Criteria:

* Known hypersensitivity or poor tolerance to bromfenac sodium or any component of the IMP or any of the procedural medications
* Currently pregnant, nursing, or planning a pregnancy; or be a woman that has a positive pregnancy test
* Currently suffer from alcohol and/or drug abuse
* Prior (within 30 days of beginning study treatment) or anticipated concurrent use of an investigational drug or device
* A condition or a situation, which in the investigator's opinion may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation
* Additional inclusion criteria also apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle: DuraSite vehicle dosed BID
Period: Overall Study
Arm/Group | ISV-303 | Vehicle
Started | 174 | 94
Safety Population | 170 | 85
mITT Population | 168 | 85
Completed | 137 | 48
Not Completed | 37 | 46

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat: subjects who were randomized into the trial, underwent cataract surgery, and received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | ISV-303 | Vehicle | Total
Number analyzed (Participants) | 168 | 85 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.90) | 72.0 (9.07) | 70.4 (9.01)
Age, Customized [Number; unit: participants]
  < 65 years | 44 | 16 | 60
  ≥ 65 years | 124 | 69 | 193
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 48 | 153
  Male | 63 | 37 | 100

OUTCOME MEASURES:

1. Primary Outcome: Ocular Inflammation
Description: Anterior chamber cell grade 0 at Day 15 measured on a 0 to 4 scale where "0" is 0 cells; "1" is 1-10 cells; "2" is 11-20 cells; "3" is 21-50 cells; "4" is > 50 cells, and no rescue medications.
Time Frame: 15 days
Population: Modified Intent-to-Treat (ITT) Population using Last Observation Carried Forward (LOCF) method.
Measure: Number; unit: participants
Arm/Group | ISV-303 | Vehicle
Number analyzed (Participants) | 168 | 85
participants | 64 | 19

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | ISV-303 | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/170 | 1/85
Other Adverse Events (participants affected / at risk) | 17/170 | 5/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-303 (N=170) | Vehicle (N=85)
Colitis (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-303 (N=170) | Vehicle (N=85)
Ocular hypertension (Eye disorders) | 17 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other